CLINICAL TRIAL: NCT03066206
Title: A Phase II Study of Poziotinib in EGFR or HER2 Mutant Advanced Solid Tumors
Brief Title: Poziotinib in EGFR Exon 20 Mutant Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0783; NCI-2017-00831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0783 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: EGFR Exon 20 Mutation; ERBB2 Gene Mutation; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (poziotinib) (Experimental): Patients receive poziotinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — Given PO
  Other Names: HM781-36B; NOV120101

SUMMARY:
This phase II trial studies how well poziotinib works in treating patients with non-small lung cancer with an EGFR or HER2 exon 20 mutation that is stage IV or has come back (recurrent). Poziotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth..

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate (ORR) to poziotinib according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in non-small cell lung cancer (NSCLC) with EGFR exon 20 mutations.

II. Assess the objective response rate (ORR) to poziotinib according to RECIST 1.1 criteria in NSCLC with HER2 (ErBB2) exon 20 mutations.

III. Assess the objective response rate (ORR) to poziotinib according to RECIST 1.1 criteria in advanced solid tumors with EGFR exon 20 or HER2 exon 20 mutations.

IV. Assess the objective response rate (ORR) to poziotinib according to RECIST 1.1 criteria in advanced solid tumors with HER2 exon 19 mutations ORR will be calculated as the percent of patients whose best confirmed response is complete response (CR, defined as disappearance of all target lesions) or partial response (PR, defined as at least a 30% decrease in the sum of longest diameter [LD] of target lesions, taking as reference the baseline sum LD).

SECONDARY OBJECTIVES:

I. Disease control rate (complete response + partial response + stable response) of poziotinb in cohort 1 and 2, analyzed independently.

II. Progression free survival of poziotinb in cohort 1 and 2, analyzed independently.

III. Overall survival of poziotinb in cohort 1 and 2, analyzed independently. IV. Duration of response of poziotinb in cohort 1 and 2, analyzed independently.

V. Safety and toxicity.

EXPLORATORY OBJECTIVES:

I. To assess molecular markers associated with resistance and response to poziotinib, including secondary mutations.

OUTLINE:

Patients receive poziotinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV or recurrent solid tumor not amenable to curative intent therapy
* Cohort 1 specific inclusion criteria: NSCLC with documented EGFR exon 20 mutation by one of the following Clinical Laboratory Improvement Act (CLIA) certified tests: OncoMine Comprehensive Assay (OCA), Guardant360 Assay (using plasma), or FoundationOne Assay or by a Food and Drug Administration (FDA) approved device using cobas EGFR mutation test version (v)2 or therascreen EGFR RGQ PCt kit; Mutations include D770_N771insSVD, D770_N771insNPG, V769_D770insASV, H773_V774insNPH, or any other exon 20 in-frame insertion or point mutation excluding T790M
* Cohort 2 specific inclusion criteria: NSCLC with documented HER2 exon 20 mutation by a CLIA certified tests: Oncomine Comprehensive Assay (OCA), Guardant360 Assay (using plasma), or FoundationOne Assay; eligible mutations include A775_G776insYVMA, G776_V777insVC, or P780_Y781insGSP, or any other in-frame exon 20 insertion mutation or point mutation including, but not limited to, L755S, G776V, and V777L
* Cohort 3 specific inclusion criteria: NSCLC with documented EGFR exon 20 mutation (excluding T790M) by one of the following CLIA certified tests: OncoMine Comprehensive Assay (OCA), Guardant360 Assay (using plasma), or FoundationOne Assay or by an FDA approved device using cobas EGFR mutation test v2 or therascreen EGFR RGQ PCt kit; mutations include D770_N771insSVD, D770_N771insNPG, V769_D770insASV, H773_V774insNPH, or any other exon 20 in-frame insertion or point mutation excluding T790M
* Cohort 4 specific inclusion criteria: solid tumor (excluding NSCLC) harboring EGFR or HER2 exon 20 mutations documented by one of the following CLIA certified tests: Oncomine Comprehensive Assay (OCA), Guardant360 Assay (using plasma), or FoundationOne Assay
* Cohort 5 specific inclusion criteria: solid tumor harboring HER2 exon 19 mutation documented by one of the following CLIA certified tests: Oncomine Comprehensive Assay (OCA), Guardant360 Assay (using plasma), or FoundationOne Assay
* Patients must have exhausted all FDA-approved standard of care options for locally advanced or metastatic disease, or are ineligible for FDA-approved standard of care options, or refusing to receive FDA-approved standard of care options. Previously untreated patients are allowed only in cohort 1 and 3 and are eligible only if EGFR Exon 20 mutation is confirmed using an FDA approved device/test such as cobas EGFR Mutation Test v2, therascreen EGFR RGQ PCR Kit or other FDA tests prior to study enrollment
* Patient has adequate tumor tissue obtained from a biopsy or surgical procedure to enable molecular profiling for retrospective central laboratory confirmation of the mutation. If tissue is not available, the patient must have biopsy accessible disease and must be willing to undergo a biopsy prior to the study
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Ability to take pills by mouth
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 institutional upper limit of normal of =< 5 x ULN if liver metastases are present
* Alkaline phosphatase =< 2.5 institutional upper limit of normal of =< 5 x ULN if liver metastases are present
* Creatinine clearance >= 50 mL/min/1.73 m^2 by Cockcroft-Gault equation
* Brain metastases are allowed, as long as they are stable and do not require treatment with anticonvulsants or escalating doses of steroids
* Females of childbearing potential must have a negative serum or urine pregnancy test and must agree to use adequate contraception for the duration of the study and six months after; adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence; females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause); women will be considered post-menopausal if they have been amenorrheic for the past 12 months without an alternative medical cause
* The following age-specific requirements must also apply:

  * Women < 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of exogenous hormonal treatments; the levels of luteinizing hormone (LH) and follicle-stimulating hormone (FSH) must also be in the post-menopausal range (as per the institution)
  * Women >= 50 years old: they would be considered post-menopausal if they have been amenorrheic for the past 12 months or more following cessation of all exogenous hormonal treatments, or have had radiation-induced oophorectomy with the last menses > 1 year ago, or have had chemotherapy-induced menopause with > 1 year interval since last menses, or have had surgical sterilization by either bilateral oophorectomy or hysterectomy
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use adequate contraception for the duration of the study and 90 days after the last dose of study medication; adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide, cervical/vault cap or intrauterine device), and abstinence
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* EGFR T790M mutation or any other acquired EGFR exon 20 mutation; patients with coexisting primary EGFR exon 20 and T790M mutations are eligible
* Have received or are receiving an investigational medicinal product (IMP) or other systemic anticancer treatment within 2 weeks prior to the first dose of study treatment
* Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment
* Have known or suspected brain metastases or spinal cord compression, unless the condition has been asymptomatic, has been treated with surgery and/or radiation, and has been stable without requiring escalating corticosteroids nor anti-convulsant medications for at least 4 weeks prior to the first dose of study medication
* Known hypersensitivity to poziotinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to poziotinib
* Cardiac conditions as follows:

  * Patient has a history of congestive heart failure (CHF) class III/IV according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment
  * Patient has a cardiac ejection fraction < 50% by either echocardiogram or multi-gated acquisition (MUGA) scan
* Have any unresolved chronic toxicity with Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade >= 2, from previous anticancer therapy, except for alopecia
* Patient is unable to take drugs orally due to disorders or diseases that may affect gastrointestinal function, such as inflammatory bowel diseases (e.g., Crohn's disease, ulcerative colitis) or malabsorption syndrome, or procedures that may affect gastrointestinal function, such as gastrectomy, enterectomy, or colectomy
* Have any condition or illness that, in the opinion of the investigator, might compromise patient safety or interfere with the evaluation of the safety of the drug
* Pregnant or breastfeeding women
* History of another primary malignancy within 2 years prior to starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ
* Recent major surgery within 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access
* Male or female patients of reproductive potential who are not employing an adequate method of birth control; adequate contraception methods include: birth control pills (e.g. combined oral contraceptive pill), barrier protection (e.g. condom plus spermicide cervical/vault cap or intrauterine device), and abstinence
* Uncontrolled intercurrent illness including, but not limited to, uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including hepatitis B, hepatitis C, human immunodeficiency virus [HIV], and active clinical tuberculosis), or renal transplant; ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements
* Active bleeding disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate a in patients with estimated glomerular filtration rate (EGFR) exon 20 mutant non-small Cell Lung Cancer (NSCLC) (Cohort 1) | Up to 4 years
  According to Response Evaluation Criteria in Solid Tumors 1.1 criteria.
Objective response rate a in patients with human epidermal growth factor receptor 2 (HER2) exon 20 mutant non-small Cell Lung Cancer (NSCLC) (Cohort 2) | Up to 4 years
  According to Response Evaluation Criteria in Solid Tumors 1.1 criteria.

SECONDARY OUTCOMES:
Disease control rate (complete response + partial response + stable disease) of poziotinb in cohort 1 and 2, analyzed independently | Up to 4 years
  Will be estimated along with 95% confidence intervals.
Progression free survival of poziotinb in cohort 1 and 2, analyzed independently | Up to 4 years
  Will be estimated using the Kaplan-Meier method and the comparison between or among patient's characteristic groups will be evaluated by log-rank test. The Cox regression model may be applied to assess the effect of covariates of interest on progression free survival.
Overall survival of poziotinb in cohort 1 and 2, analyzed independently | Up to 4 years
  Will be estimated using the Kaplan-Meier method and the comparison between or among patient's characteristic groups will be evaluated by log-rank test. The Cox regression model may be applied to assess the effect of covariates of interest on overall survival.
Duration of response of poziotinb in cohort 1 and 2, analyzed independently | Up to 4 years
  Duration of response will be measured.
Incidence of adverse events | Up to 4 years
  Assessed by Common Terminology Criteria for Adverse Events version 4.03. Toxicity data will be summarized by frequency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Y Elamin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Elamin YY, Robichaux JP, Carter BW, Altan M, Tran H, Gibbons DL, Heeke S, Fossella FV, Lam VK, Le X, Negrao MV, Nilsson MB, Patel A, Vijayan RSK, Cross JB, Zhang J, Byers LA, Lu C, Cascone T, Feng L, Luthra R, San Lucas FA, Mantha G, Routbort M, Blumenschein G Jr, Tsao AS, Heymach JV. Poziotinib for EGFR exon 20-mutant NSCLC: Clinical efficacy, resistance mechanisms, and impact of insertion location on drug sensitivity. Cancer Cell. 2022 Jul 11;40(7):754-767.e6. doi: 10.1016/j.ccell.2022.06.006. PMID 35820397
- [Derived] Elamin YY, Robichaux JP, Carter BW, Altan M, Gibbons DL, Fossella FV, Lam VK, Patel AB, Negrao MV, Le X, Mott FE, Zhang J, Feng L, Blumenschein G Jr, Tsao AS, Heymach JV. Poziotinib for Patients With HER2 Exon 20 Mutant Non-Small-Cell Lung Cancer: Results From a Phase II Trial. J Clin Oncol. 2022 Mar 1;40(7):702-709. doi: 10.1200/JCO.21.01113. Epub 2021 Sep 22. PMID 34550757
- See also: MD Anderson Cancer Center — http://www.mdanderson.org